CLINICAL TRIAL: NCT05822154
Title: Comprehensive Geriatric Assessment in the Elderly Subjects (PROMISING)
Acronym: PROMISING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: INRCA_001_2023
Record Dates: First submitted 2023-03-27; First posted 2023-04-20 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-03

CONDITIONS: Ageing; Frailty
Keywords: ageing; comprehensive geriatric assessment; polypharmacy
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly subjects: subjects aged 65 years and over
  Interventions: Other: comprehensive geriatric assessment

INTERVENTIONS:
Other: comprehensive geriatric assessment — The clinical, biological and functional characteristics will be collected in elderly subjects attending the hospitals of participating centers.

SUMMARY:
The primary objective of this observational study is to verify, through a comprehensive geriatric assessment, the health status of a sample of elderly subjects.

DETAILED DESCRIPTION:
The primary objective of this observational study is to verify, through a comprehensive geriatric assessment, the health status of a sample of elderly subjects. Short- to medium-term outcomes will also be evaluated through follow-up.

ELIGIBILITY:
Inclusion Criteria:

* subjects with 65 years or older

Exclusion Criteria:

* no informed consent

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients from different settings (inpatients and outpatients) who attend the hospitals of the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in health conditions | Baseline, 3, 6 and 12 months later
  The prevalence of comorbidities and their risk factors at time of enrolment
Change in prevalence of polypharmacy | Baseline, 3, 6 and 12 months later
  Number of participants with polypharmacy. Polypharmacy will be defined as being on five or more medications at one time

SECONDARY OUTCOMES:
Change in frailty condition | Baseline, 3, 6 and 12 months later
  Clinical Frailty Scale (CFS). The CFS divides patients into 9 classes from very fit (CFS=1) to terminally ill (CFS=9)
Change in functional capacity | Baseline, 3, 6 and 12 months later
  Activity of Daily Living (ADL). A summary score ranges from 0 (low function, dependent) to 6 (high function, independent)
Change in functional capacity | Baseline, 3, 6 and 12 months later
  Activity of Instrumental of Daily Living (IADL). A summary score ranges from 0 (low function, dependent) to 8 (high function, independent)
Change in physical performance | Baseline, 3, 6 and 12 months later
  Physical performance will be ascertained using the Short Physical Performance Battery (SPPB). Summary scores range from 0-12 and higher scores denote higher physical performance
Change of cognitive function score | Baseline, 3, 6 and 12 months late
  Mini-mental State Examination (0-30 points), the higher the score, the better the cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Corsonello, MD, Principal Investigator — IRCCS INRCA, Cosenza, Italy; Simona Ciccone, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano, Italy; Antonio Greco, MD, Principal Investigator — Casa Sollievo della Sofferenza, San Giovanni Rotondo, Italy; Rodolfo Sardone, MD, Principal Investigator — IRCCS "Saverio de Bellis", Castellana Grotte (BA), Italy; Fabrizio Giunco, MD, Principal Investigator — Fondazione Don Carlo Gnocchi, Milano, Italy; Mariacristina Parravano, MD, Principal Investigator — Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia, Roma, Italy; Marco Lenti, MD, Principal Investigator — Fondazione Policlinico San Matteo, Pavia, Italy; Rosa Liperoti, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, Roma, Italy; Francesca Bruni, MD, Principal Investigator — Istituto Auxologico Italiano, Milano, Italy; Giuseppe Rengo, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri, Scientific Institute of Telese Terme (BN), Italy; Milena Fini, MD, Principal Investigator — Istituto Ortopedico Rizzoli, Bologna, Italy; Luigi Zagra, MD, Principal Investigator — Istituto Ortopedico Galeazzi, Milano, Italy; Alessandro Nobili, MD, Principal Investigator — Istituto di Ricerche Farmacologiche Mario Negri, Milano, Italy
Locations (1):
- IRCCS INRCA Hospital, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: No